CLINICAL TRIAL: NCT05126368
Title: Rotational Stability of the TECNIS Eyhance Toric II IOL
Brief Title: Rotational Stability of the TECNIS Eyhance Toric
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eyhance Toric
Record Dates: First submitted 2021-11-02; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cataract
Keywords: Cataract; Astigmatism; Toric intraocular lens
MeSH Terms: conditions — Cataract; Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyhance toric II (Experimental): The Eyhance toric II intraocular lens will be implanted in one of the patients eyes during cataract surgery
  Interventions: Other: Cataract surgery

INTERVENTIONS:
Other: Cataract surgery — During cataract surgery the Eyhance toric II intraocular lens will be implanted in one eye of the patient

SUMMARY:
Evaluation of the rotational stability of a new toric intraocular lens (IOL), the TECNIS Eyhance toric II.

DETAILED DESCRIPTION:
With increasing demands of patients concerning the refractive outcome after cataract surgery, toric intraocular lenses (IOLs) have become more popular. Originally, toric IOLs were used mainly to correct corneal astigmatism in patients with high degrees of astigmatism. Since a couple of years, toric IOLs are available from numerous manufacturers to correct moderate or even low amounts of astigmatism which are much more prevalent. Only about 8% of the population has a corneal astigmatism of 2.0 D or more, while the incidence of a corneal astigmatism of 0.75 D or more is about 30%. The use of toric IOLs in this population results in less spectacle dependence due to the astigmatic correction.

Toric IOLs became the gold standard to correct corneal astigmatism during cataract surgery and rotational stability and axis alignment are critical to the efficacy of the surgical outcome. Misalignment may be caused intra- or postoperatively. Intraoperatively, misalignment may happen due to cyclotorsion of the eye in supine position or due to peribulbar anaesthesia and imprecision of positioning the IOL along the correct meridian in the capsular bag. This can be compensated for by preoperative corneal marking in the sitting position and meticulous positioning of the IOL during surgery. However, there are several other risk factors that influence rotational stability in the postoperative period, such as IOL design, haptic design and material, axial length, capsulorhexis size, capsular bag diameter and capsular bag shrinkage.

Long-term success of toric IOLs depends on rotational stability, nevertheless rotation mostly happens in the early postoperative period and once the anterior and posterior capsules fuse, IOL rotation is less frequent. A study by Kim et al. showed no significant differences in lens rotation between the early and late postoperative follow-up, and Kwartz et al. showed no significant differences between the two periods when different lens materials were used. Varsits et al. reported that rotation of toric IOLs is typically seen within the first hour after implantation.

It is known that tilt and decentration of the IOL can lead to a negative effect on optical performance and horizontal tilt induces against-the-rule-astigmatism. Every degree of rotation results in a loss of 3.3% of cylindrical power and misalignment of more than 10 degrees is considered an indication of surgical repositioning.

The aim of this study is therefore to evaluate the rotational stability of the TECNIS Eyhance toric II intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Age 21 and older
* Regular corneal astigmatism > 0.75 dioptres
* Written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation, traumatic cataract, corneal scars or other co-morbidities that could affect capsular bag stability (e.g. Marfan syndrome)
* High myopia (> 29 mm AL)
* Irregular corneal astigmatism on corneal topography
* Pregnancy (a pregnancy test will be taken preoperatively in women of reproductive age)

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-04-29 (Estimated); Study Completion 2022-11-29 (Estimated)

PRIMARY OUTCOMES:
Rotational stability | 12 months
  The change in the intraocular lens axis (given in degrees) of the Eyhance toric IOL of one eye will be analysed by taking photographs of the IOL and will be compared between the different study time points.

SECONDARY OUTCOMES:
Distance visual acuity | 12 months
  Distance visual acuity will be determined using ETDRS-charts in a distance of 4 metres and differences in refraction will be compared between the different study time points.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zeilinger J, Hienert J, Ruiss M, Pilwachs C, Findl O. Rotational stability of a new toric intraocular lens with an advanced optical profile. J Cataract Refract Surg. 2023 Jun 1;49(6):584-588. doi: 10.1097/j.jcrs.0000000000001158. PMID 36745852